CLINICAL TRIAL: NCT01266239
Title: Japanese Registry Study in Comparison Between Everolimus-eluting Stent and Sirolimus-eluting Stent for the Bifurcation Lesion
Brief Title: Comparison Between Everolimus-eluting Stent (EES) and Sirolimus-eluting Stent (SES) in the Bifurcation Lesion
Acronym: J-REVERSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Yukuhashi Hospital (Network)
Collaborators: Abbott Medical Devices (Industry); Cordis US Corp. (Industry)
Responsible Party: Yoshinobu Murasato, New Yukuhashi Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: J-REVERSE
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Ischemic Heart Disease
Keywords: Bifurcation lesion, drug-eluting stent, symmetric expansion
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SES-KB (Active Comparator): Sirolimus-eluting stent (SES) is deployed in the main vessel (MV)and subsequent kissing balloon inflation is performed in the bifurcation.
  Interventions: Procedure: kissing balloon inflation; Device: EES vs. SES
- SES-NK (Active Comparator): SES is deployed in the MV without kissing balloon inflation.
  Interventions: Procedure: kissing balloon inflation; Device: EES vs. SES
- EES-KB (Active Comparator): Everolimus-eluting stent (EES) is deployed in the MV and subsequent kissing balloon inflation is performed in the bifurcation.
  Interventions: Procedure: kissing balloon inflation; Device: EES vs. SES
- EES-NK (Active Comparator): EES is deployed in the MV without kissing balloon inflation.
  Interventions: Procedure: kissing balloon inflation; Device: EES vs. SES

INTERVENTIONS:
Procedure: kissing balloon inflation — Kissing balloon inflation following the MV stenting
Device: EES vs. SES — Rapid endothelialization after EES deployment has been reported compared to that after SES deployment.

SUMMARY:
In study-1, the purpose of this study is to compare the long-term outcome of provisional stenting between EES and SES deployment. In study-2, it is to prove the following hypothesis " Asymmetrical expansion in the bifurcation lesion leads to frequent inhomogeneous intimal growth on the strut and thrombus attachment."

DETAILED DESCRIPTION:
Kissing balloon inflation brings asymmetrical expansion which may lead to a risk of disturbance of endothelialization. We will investigate the following issues.

1. Impact of asymmetric expansion induced by kissing balloon technique on mid and long term results
2. Difference between SES and EES
3. Impact of abnormal OCT findings on long-term clinical outcome (3yr)

ELIGIBILITY:
Inclusion Criteria:

1. Coronary bifurcation lesion which stenotic lesion exists in the MV and / or in the side branch (SB).
2. The lesion is appropriate for the provisional MV stenting.
3. The reference diameter is more than 2.5mm in the MV and more than 2.0mm in the SB.

Exclusion Criteria:

1. Left main coronary bifurcation
2. Acute myocardial infarction and unstable angina which culprit vessel contains obvious thrombus
3. Left ventricular ejection fraction < 30%
4. Shock state
5. Inappropriate candidate for the dual antiplatelet therapy, administration of contrast medium and radiation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 3 years
  Cardiac death, myocardila infarction, target lesion revascularization, target vessel revascularization, and stent thrombosis are monitored.

SECONDARY OUTCOMES:
abnormal intimal coverage | 9 months
  Optical coherence tomography (OCT) is planned at the 9-month follow-up period. Unevenness of intimal growth, number of uncovered struts, and frequency of thrombus attachment are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshinobu Murasato, MD, PhD, Principal Investigator — New Yukuhashi Hospital; Yoshihisa Kinoshita, MD, Principal Investigator — Toyohashi Heart Center
Locations (5):
- Japan (5):
  - Kobe University, Kobe
  - Hyogo Medical University, Nishinomiya
  - Toyohashi Heart Center, Toyohashi
  - Saiseikai Yokohama Eastern Hospital, Yokohama
  - New Yukuhashi hospital, Yukuhashi